CLINICAL TRIAL: NCT05479955
Title: The Effect of Skin to Skin Contact Time After Childbirth on Fear of Child Birth, Birth Trauma and Maternal Attachment: A Single-blind Randomized Controlled Trial
Brief Title: Skin-to-skin Contact Time and Maternal Psychology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gozde Gokce Isbir, Associate Prof, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GGI
Record Dates: First submitted 2022-07-15; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Skin to Skin Contact

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 minutes skin to skin contact (Experimental): Participants were provided care in different rooms, blinded to the differences in practice used between the two groups. Skin-to-skin contact was applied to the babies of the women in this group for 5 minutes immediately after birth. After the application, routine follow-up and care of the newborn was performed and kept under a radiant heater. When the woman became stable, her baby was given and breastfeeding was supported.
  Interventions: Other: 5 minutes skin to skin contact
- 60 minutes skin to skin contact (Experimental): Participants were provided care in different rooms, blinded to the differences in practice used between the two groups. Skin-to-skin contact application was initiated to the babies of the women in this group immediately after birth and was applied continuously for 60 minutes as recommended by WHO. Follow-up and care of the newborn were done during the application. At the end of 60 minutes, the baby was dressed and given to its mother.
  Interventions: Other: 60 minutes skin to skin contact

INTERVENTIONS:
Other: 5 minutes skin to skin contact — Skin-to-skin contact is defined as placing a naked baby on the mother's bare stomach or breast for at least one hour immediately after birth. The women in this group received 5 minutes of skin-to-skin contact as a clinic routine.
  Arms: 5 minutes skin to skin contact
Other: 60 minutes skin to skin contact — Skin-to-skin contact is defined as placing a naked baby on the mother's bare stomach or breast for at least one hour immediately after birth. In line with the recommendation of the World Health Organization, 60 minutes of skin-to-skin contact was applied to the women in this group.
  Arms: 60 minutes skin to skin contact

SUMMARY:
The aim of this study was to determine the effect of postpartum skin-to-skin contact time on fear of childbirth, birth trauma and maternal attachment.

DETAILED DESCRIPTION:
This is a single-blind, randomized controlled trial. Data were collected from 110 women who gave birth in the gynecology clinic of a public hospital in southern Turkey between September 2021 and February 2022. Participants who met the inclusion criteria were informed about the purpose of the study and skin-to-skin contact, informed consent was obtained from those who agreed to participate, and the women were divided into groups according to a 1:1 computer-based randomization program. Data were collected at the time of consent to the study, within the first hour after birth, 24 hours after birth, 4 weeks postpartum, and 4 months postpartum. Collected by the first author. The CONSORT directive was followed in the planning, implementation and writing of the research.

ELIGIBILITY:
Inclusion Criteria

* Must be able to a normal term vaginal delivery,
* Native language is Turkish,
* Have single fetus
* Must be able to skin to skin contact wit her baby

Exclusion Criteria

* Cesarean section,
* Complications,
* Psychological or psychiatric disorder,

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Level of Fear of Childbirth | Postpartum with in 4th- 24th hours
  Women's fears after childbirth were evaluated with the Wijma Delivery Expectancy/Experience Questionnaire Version B version (W-DEQ-B).
  This scale was developed by Wijma et al (1998) for fear after childbirth. The Turkish validity and reliability of the scale were performed by Korukcu et al. (2016). This scale consisting of 33 items is a 5-point Likert-type. The positive-meaning items are scored in reverse order. Therefore, the scores ranged from 0 to 165. The scale has no cutoff score, and high scores indicated higher fear.
Level of Birth Trauma | Postpartum 4th weeks
  Birth trauma of women were evaluated with the City Birth Trauma Scale. City BiTS was developed by Ayers et al., (2018) to measure birth trauma. The Turkish validity and reliability of the scale were performed by Bayrı Bingöl et al. (2021). The scale is a fourpoint Likert-type instrument composed of 29 items. Higher scores reflect greater risk for Post-traumatic Stress Disorder (PTSD). The Cronbach's alpha for the original scale was measured as .92 (Ayers et al.,2018) and Turkish version was measured as 0.91 (Bayrı Bingöl et al., 2021). In this study, 6-8 days after birth to determine whether they meet the criteria for birth trauma and birth-related PTSD.
Level of Maternal Attachment | Postpartum 4th weeks
  Maternal attachment of women was evaluated with the Maternal Attachment Inventory.
  MAI, was developed by Muller (1994) to measure maternal attachment. The Turkish validity and reliability of the scale were performed by Kavlak et al. (2009). This scale consisting of 26 items is a 4-point Likert-type (4 = every time to 1 = any time). The scores ranged from 26 to 104 and high scores indicated higher maternal attachment. The Cronbach's alpha for the original scale was measured as .76 - .85 at different time (Muller, 1994) and Turkish version was measured as 0.77 (Kavlak et al., 2009). In this study, 6th to 8th postnatal days were used to measure maternal attachment.
Level of Birth Trauma | Postpartum 4th month
  Birth trauma of women were evaluated with the City Birth Trauma Scale. City BiTS was developed by Ayers et al., (2018) to measure birth trauma. The Turkish validity and reliability of the scale were performed by Bayrı Bingöl et al. (2021). The scale is a fourpoint Likert-type instrument composed of 29 items. Higher scores reflect greater risk for Post-traumatic Stress Disorder (PTSD). The Cronbach's alpha for the original scale was measured as .92 (Ayers et al.,2018) and Turkish version was measured as 0.91 (Bayrı Bingöl et al., 2021). In this study, 6-8 days after birth to determine whether they meet the criteria for birth trauma and birth-related PTSD.
Level of Maternal Attachment | Postpartum 4th month
  Maternal attachment of women was evaluated with the Maternal Attachment Inventory.
  MAI, was developed by Muller (1994) to measure maternal attachment. The Turkish validity and reliability of the scale were performed by Kavlak et al. (2009). This scale consisting of 26 items is a 4-point Likert-type (4 = every time to 1 = any time). The scores ranged from 26 to 104 and high scores indicated higher maternal attachment. The Cronbach's alpha for the original scale was measured as .76 - .85 at different time (Muller, 1994) and Turkish version was measured as 0.77 (Kavlak et al., 2009). In this study, 6th to 8th postnatal days were used to measure maternal attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Gozde Gokce Isbir, Principal Investigator — Mersin University
Locations (1):
- Gozde Gokce Isbir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No